CLINICAL TRIAL: NCT01237977
Title: Double-blind, Randomized, Active Drug Comparative, Parallel Designed, Multi-center,Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of "Meditoxin® Versus Botox® in the Treatment of Glabellar Lines
Brief Title: Efficacy and Safety Study of Botulinum Toxin Type A to Treat Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSP-MDTX-GL-0901
Record Dates: First submitted 2010-11-04; First posted 2010-11-10 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Skin Aging
MeSH Terms: interventions — Botulinum Toxins, Type A; 3-deoxyglycero-galacto-nonulosonic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin type A(Meditoxin®) (Experimental)
  Interventions: Drug: Botulinum Toxin Type A(Meditoxin®)
- Botulinum toxin type A(Botox®) (Active Comparator)
  Interventions: Drug: Botulinum Toxin Type A(Botox®)

INTERVENTIONS:
Drug: Botulinum Toxin Type A(Meditoxin®) — single administration, Day 0, 20U
  Other Names: Neuronox®, Siax®
  Arms: Botulinum toxin type A(Meditoxin®)
Drug: Botulinum Toxin Type A(Botox®) — single administration, Day 0, 20U
  Arms: Botulinum toxin type A(Botox®)

SUMMARY:
The purpose of this study is to test the hypothesis that the efficacy and safety of Meditoxin® are not inferior to Botox®'s in the treatment of glabellar lines.

DETAILED DESCRIPTION:
The allocated subject is injected Investigational Product(Meditoxin® or Botox®) 20U in middle of the forehead. The efficacy and safety are evaluated for 16weeks through 4 follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 20 and 65
* Patients attaining ≥grade 2 (moderate) in the investigator's rating of the severity of glabella lines at maximum frown
* Patients who can comply with the study procedures and visit schedule
* Patients who voluntarily sign the informed consent

Exclusion Criteria:

* Patients with medical conditions who may be at greater risk due to the administration of the investigational drugs (e.g.. diseases that may affect the neuromuscular action including Myasthenia Gravis, Lambert-Eaton Syndrome, Amyotrophic Lateral Sclerosis and motor neuropathy)
* Patients with severe internal diseases (cardiovascular, respiratory, endocrine diseases etc.)
* Patients who have bleeding tendency or taking anti-coagulant
* Patients who were injected with botulinum toxin within the past 3 months
* Patients with allergy or hypersensitivity to the investigational drugs or their components
* Female subjects who are pregnant or lactating. Female subjects of childbearing age who have a plan to get pregnant during the study period, or do not use available contraceptive methods (Women of childbearing age should have negative urine pregnancy test results at baseline visit (0 week) prior to the first injection.)
* Patients with the history of facial nerve paralysis or the symptoms of eyelid ptosis
* Patients with skin disorders or infection at the injection site
* Patients who have received other procedures which may affect glabellar and forehead lines within 6 months
* Patients with the history of treatment of glabellar part(including forehead) like face lifting and permanent implant or with scars which may affect the treatment results
* Patients whose glabellar lines cannot be satisfactorily improved with physical method since the lines are not flattened even using hands
* Patients who have a plan to receive facial cosmetic procedures including dermal filler, photorejuvenation, chemical peeling and dermabrasion during the study period
* Patients who are participating in other clinical trials or have participated in other clinical trials 30 days before screening or the five times the half life of a drug which was given to patient during the previous clinical trials
* Patients who are unable to communicate or follow the instructions
* Patients who are not eligible for this study based on the judgment of an investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2009-11-23 (Actual); Primary Completion 2010-08-30 (Actual); Study Completion 2010-09-30 (Actual)

PRIMARY OUTCOMES:
Glabellar line improvement rate at maximum frown confirmed with investigator's live assessment severity | 0 and 4 weeks after the injection
  Glabellar line improvement rate at maximum frown confirmed with investigator's live assessment of glabellar line severity at baseline and 4 weeks after the injection

SECONDARY OUTCOMES:
Glabellar line improvement rate at maximum frown confirmed with investigator's live assessment | 0, 8, 12 and 16 weeks after the injection
  Glabellar line improvement rate at maximum frown confirmed with investigator's live assessment at baseline, 8, 12 and 16 weeks after the injection
Glabellar line improvement rate at rest confirmed with investigator's live assessment of glabellar line severity | 0, 4, 8, 12 and 16 weeks after the injection
  Glabellar line improvement rate at rest confirmed with investigator's live assessment of glabellar line severity at baseline, 4, 8, 12 and 16 weeks after the injection
Glabellar line improvement rate at maximum frown confirmed with investigator's photo assessment | 0, 4, 8,12 and 16 weeks after the injection
  Glabellar line improvement rate at maximum frown confirmed with investigator's photo assessment at baseline, 4, 8,12, 16 weeks after the injection
Glabellar line improvement rate at rest confirmed with investigator's photo assessment of glabellar line severity | 0, 4, 8, 12 and 16 weeks after the injection
  Glabellar line improvement rate at rest confirmed with investigator's photo assessment of glabellar line severity at baseline, 4, 8, 12 and 16 weeks after the injection
Glabellar line improvement rate confirmed with subject's assessment | 4, 8, 12 and 16 weeks after the injection
  Glabellar line improvement rate confirmed with subject's assessment at 4, 8, 12 and 16 weeks after the injection
Subject satisfaction rate | 4, 8, 12 and 16 weeks after the injection
  Subject satisfaction rate at 4, 8, 12 and 16 weeks after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hun Huh, MD, Ph.D., Principal Investigator — Seoul National University Bundang Hospital; Hoon Kang, MD, Ph.D., Principal Investigator — St. Paul Hospital; Won-Seok Kim, MD, Ph.D., Principal Investigator — Kang-Buk Samsung Medical Center; Jong-Hyun Won, MD, Ph.D., Principal Investigator — Seoul Asan Medical Center; Joo-Hee Lee, MD, Ph.D., Principal Investigator — Sevrance Medical Center; Beom-Joon Kim, MD, Ph.D., Principal Investigator — Chung-Ang University Yong-San Hospital
Locations (6):
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyoung-gi Do
  - Kangbuk Samsung Medical Center, Seoul
  - Sevrance Medical Center, Seoul
  - St. Paul Hospital, Seoul
  - Seoul Asan Medical Center, Seoul
  - Chung-Ang University Yong-San Hospital, Seoul

REFERENCES:
- [Result] Carruthers JD, Lowe NJ, Menter MA, Gibson J, Eadie N; Botox Glabellar Lines II Study Group. Double-blind, placebo-controlled study of the safety and efficacy of botulinum toxin type A for patients with glabellar lines. Plast Reconstr Surg. 2003 Sep 15;112(4):1089-98. doi: 10.1097/01.PRS.0000076504.79727.62. PMID 12973229
- [Result] Kriegl L, Horst D, Kirchner T, Jung A. LEF-1 expression in basal cell carcinomas. Br J Dermatol. 2009 Jun;160(6):1353-6. doi: 10.1111/j.1365-2133.2009.09144.x. Epub 2009 Mar 30. No abstract available. PMID 19416246
- [Result] Walter SD, Eliasziw M, Donner A. Sample size and optimal designs for reliability studies. Stat Med. 1998 Jan 15;17(1):101-10. doi: 10.1002/(sici)1097-0258(19980115)17:13.0.co;2-e. PMID 9463853
- [Result] Landis JR, Koch GG. An application of hierarchical kappa-type statistics in the assessment of majority agreement among multiple observers. Biometrics. 1977 Jun;33(2):363-74. No abstract available. PMID 884196